CLINICAL TRIAL: NCT01694511
Title: High Resolution Magnifying Endoscopy and Contrast Enhanced Imaging Versus Standard White Light Endoscopy for the Detection of Dysplasia in Barrett's Esophagus. A Prospective Blinded Cross-over Study.
Brief Title: Endoscopic Detection of Dysplasia in Barrett's Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2-2188
Record Dates: First submitted 2012-09-17; First posted 2012-09-27 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Barrett's Esophagus
Keywords: Endoscopy, Gastrointestinal
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Introductory conventional endoscopy (Active Comparator): Conventional endoscopy followed by HRME+CVC after 30 days.
  Interventions: Procedure: HRME+CVC
- Introductory HRME+CVC (Active Comparator): HRME+CVC followed by conventional endoscopy after 30 days.
  Interventions: Procedure: conventional endoscopy

INTERVENTIONS:
Procedure: HRME+CVC — High resolution magnification endoscopy with computed virtual chromoendoscopy and directed biopsy
  Arms: Introductory conventional endoscopy
Procedure: conventional endoscopy — Conventional white light endoscopy with four-quadrant biopsy
  Arms: Introductory HRME+CVC

SUMMARY:
The purpose of this study is to determine whether High Resolution Magnification Endoscopy (HRME) and Computed Virtual Chromoendoscopy (CVC) with targeted biopsies is superior to conventional white light endoscopy (WLE) with 4 quadrant biopsies of the metaplastic epithelium every 1-2 cm (Seattle Protocol) for detection of pre-malignant lesions in patients with Barrett's Esophagus (BE).

DETAILED DESCRIPTION:
BE is a metaplastic mucosal transformation adjacent to the esophagogastric junction, due to chronic reflux of gastric juices, Gastro Esophageal Reflux Disease (GERD). The continuous esophageal exposure of acid- and/or bile- containing fluids leads, untreated, to chronic esophagitis. In certain patients a mucosal transformation takes place. The epithelium in the distal part of esophagus is transferred from squamous into a more intestinal-like mucosa, called Specialized Intestinal Metaplasia (SIM).Patients with BE is believed to run a higher risk of developing esophageal adenocarcinoma (EAC).

EAC is a rare condition in the western society, but the prevalence is rising compared with other malignancies, and a substantial increase has been seen during the last four decades. The pathogenesis of cancer development is believed to be that SIM in some patients can undergo dysplastic transformation, from low to high grade, and from high grade dysplasia (HGD) develop into AC. Advanced EAC is associated to a poor prognosis whereas HGD or carcinoma in situ may be treated endoscopically with a favorable outcome.

The need for surveillance endoscopy in order to discover early cancer lesions available to curable treatment is up against cost effectiveness and evidence level regarding screening. The conventional endoscopic (CE) surveillance algorithm for BE is standard WLE and 4 quadrant biopsies of the metaplastic epithelium every 1-2 cm above the esophagogastric junction. The development of advanced endoscopic techniques have made it possible to distinguish minimal polypoid lesions but also the microvasculature and pit-pattern structures that in certain grading systems have been associated to presence of dysplasia. Attempts have been made in exploring the benefits of advanced endoscopic technologies against standard WLE. Feasibility-studies suggests that the new techniques improves the biopsy-yield for dysplasia, however only a limited number of prospective studies exist.

Study aim: To determine whether HRME and CVC with targeted biopsies is superior to conventional WLE with 4 quadrant biopsies of the metaplastic epithelium every 1-2 cm (Seattle Protocol) for detection of pre-malignant lesions in patients with BE.

Primary endpoint: Incidence of detected dysplasia by each endoscopic technique. Secondary endpoints: 1.The yield of low- and/or high-grade dysplasia by each endoscopic technique. 2.The number of biopsies taken and the duration of the different endoscopic techniques. 3.The endoscopic prediction capability of present dysplasia compared to histopathology for HRME.

Statistical power: Based on the primary endpoint, the amount of dysplasia in a Barrett-population is approximately 10%. We calculated a raise in positive yield with using advanced endoscopy to 8%. At p<0,05 and a power of 80% the need for 105 patients.

Setting: Tertiary referral high volume endoscopy center at Sahlgrenska University Hospital, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Presence of specialized intestinal metaplasia in biopsies from the esophagus

Exclusion Criteria:

* Dysplasia or cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Incidence of detected dysplasia by each endoscopic technique. | Up to 36 months.

SECONDARY OUTCOMES:
The yield of low- and/or high-grade dysplasia by each endoscopic technique. | Up to 36 months.
The number of biopsies taken and the duration of the different endoscopic techniques. | Up to 36 months.

OTHER OUTCOMES:
The endoscopic prediction capability of present dysplasia compared to histopathology for HRME. | Up to 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Anders F Edebo, MD, PhD, Study Director — Dept. Gastrosurgical Research and Education, Inst. Clinical Sciences, Sahlgrenska Academy, Gothenburg, Sweden
Locations (1):
- Gastrointestinal Endoscopy Unit, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Bratlie SO, Johnsson E, Jonsson C, Fandriks L, Edebo A. Multiple-Band Imaging Provides Better Value Than White-light Endoscopy in Detection of Dysplasia in Patients With Barrett's Esophagus. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1068-74.e2. doi: 10.1016/j.cgh.2014.12.007. Epub 2014 Dec 11. PMID 25499989